CLINICAL TRIAL: NCT06050213
Title: Maxillary Overdenture Retained by Different Number of Implants Opposed by 2-implant Assisted Mandibular Overdenture. A Cross-over Study of Patient Satisfaction
Brief Title: Edentulous Maxilla Opposed by 2-implant Mandibular Overdenture?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A20080622
Record Dates: First submitted 2023-09-17; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Prosthesis Durability
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- three implant group (Active Comparator): Maxillary overdenture retained by 3 unsplinted implants in midline and canines regions.
  Interventions: Device: Maxillary implant overdenture
- five implant group (Active Comparator): Maxillary overdenture retained by 5 unsplinted implants in midline, canines and molar regions.
  Interventions: Device: Maxillary implant overdenture
- four implant group (Active Comparator): Maxillary overdenture retained by 4 unsplinted implants in canines and molar regions.
  Interventions: Device: Maxillary implant overdenture

INTERVENTIONS:
Device: Maxillary implant overdenture — maxillary overdenture retained by different number of implants

SUMMARY:
This within -subject study will be conducted to evaluate the proper number of unsplinted implants ;( three, four and five implants) for the edentulous maxilla opposed by mandibular two-implant overdentures.

ELIGIBILITY:
Inclusion Criteria:

* o Healthy and free from any systemic diseases that may interfere with the osseointegration of implants.

  * Patients have completely edentulous maxilla for at least 6 months after last extraction with opposing mandibular two-implant Overdentures.
  * The patients have angle class I maxillomandibular skeletal relation and sufficient interarch space not less than (10-12 mm) as detected by tentative jaw relation.
  * Maxillary and mandibular alveolar ridges covered with healthy, firm, relatively even thickness and even compressible mucosa as detected by palpation with the blunt end of the mirror and free from any signs of inflammation or flabbiness as detected by clinical examination.
  * Good quality and quantity of maxillary residual alveolar ridge, as detected by CBCT, available for implant width (3.7mm, 5mm for anterior and posterior implants respectively) and length (12mm, 10mm for anterior and posterior implants respectively) this was ascertained by CBCT.

Exclusion Criteria:

* o Any history of metabolic or systemic diseases that may affect integration of implant or connective tissue health surrounding implant.

  * History of irradiation in head-and-neck area.
  * Heavy smokers (more than 10 cigarettes per day)
  * Parafunctional habits such as bruxism.
  * Psychiatric disorders or unrealistic expectations.
  * Positive pregnancy test up to 5 days before surgery.
  * Severe thrombocytopenia and bleeding disorders.
  * Pathologic condition of soft tissue (bacterial and viral stomatitis, hyperplasia, cyst, fibrous lesions)
  * Patients with local contraindications for implant placement due to localized bone defects and poor bone quality (D5).
  * Patients with TMJ disorders or poor neuromuscular coordination.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-12-26 (Estimated); Study Completion 2024-07-16 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | one year
  patient satisfaction will be evaluated for all patients by a questionnaire using visual analogue scale
Bite force | one year
  Bite force will be evaluated for all patients by a digital bite force device

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No